CLINICAL TRIAL: NCT00285909
Title: Effect of Moderate Alcohol Consumption on PPAR-γ Activity and Risk Markers of Metabolic Disease: Influence of Genetic Variation in Alcohol Oxidation
Brief Title: Moderate Alcohol Consumption, Risk of Cardiovascular Disease and Type 2 Diabetes: Influence of Alcohol Oxidation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TNO (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: P6689; Alcohol research 20
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2006-08-16 (Estimated); Status verified 2006-08

CONDITIONS: Cardiovascular Disease; Type 2 Diabetes
Keywords: Moderate alcohol consumption; Alcohol dehydrogenase 1c polymorphism; PPAR-gamma activated gene expression
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2 | interventions — Ethanol

INTERVENTIONS:
Behavioral: Alcohol: 25 gday (white wine)

SUMMARY:
Moderate alcohol consumption is associated with a decreased risk of cardiovascular disease and type 2 diabetes. The association of alcohol consumption with cardiovascular disease is mediated by a functional polymorphism of alcohol dehydrogenase 1c, but the effect of this polymorphism on alcohol metabolism is only investigated in vitro.

The risk reduction of moderate alcohol consumption for cardiovascular disease is explained largely by an increase of HDL cholesterol, but an increase of adiponectin concentrations after moderate alcohol consumption may also be involved. It seems likely that adiponectin is a mediator for the association of moderate alcohol consumption with type 2 diabetes. The mechanism by which moderate alcohol consumption increases adiponectin concentrations is unknown, but ppar-gamma activation may be involved.

effects of this polymorphism on mediators of this relation are not known. This study therefore investigates the effect of moderate alcohol consumption and the influence of alcohol dehydrogenase 1c polymorphism on ppar-gamma activated gene expression and risk factors of cardiovascular disease and type 2 diabetes.

DETAILED DESCRIPTION:
Objectives :

To investigate the effect of moderate alcohol consumption and influence of genetic variation of ethanol oxidation on:

* PPAR-γ activated gene expression
* Markers of coronary heart disease or type 2 diabetes
* Postprandial changes of HPA-axis activity among 36 postmenopausal women with ADH1C genotype associated with slow or fast alcohol metabolism.

Design : Randomized, controlled, not blinded crossover trial with 1 week wash-out preceding each treatment period

Participants

* Description : Apparently healthy postmenopausal women
* Number : 36

Study substances

* Test substance : White wine (ca. 25 g alcohol/day)
* Reference substance : White grape juice

Study treatments Treatment A: 250 ml white wine daily (ca. 25 g alcohol/day) Treatment B: 250 ml white grape juice daily

Study period

- Duration : two periods of 6 weeks preceded by 1 week wash-out period

Test parameters:

* Adiponectin mRNA expression
* Expression of PPAR-gamma activated genes: CD36, lipoprotein lipase, AP2
* Markers of cardiovascular disease (blood lipid profile, Lp-PLA2 activity, hs-CRP, fibrinogen)
* Markers of type 2 diabetes (adiponectin, adiponectin oligomers, insulin sensitivity)
* Parameters of alcohol oxidation (postprandial: blood alcohol and acetate, acetaldehyde)
* HPA-axis activity (postprandial & fasting: cortisol, ACTH, testosterone)

ELIGIBILITY:
Inclusion Criteria:

* Healthy women aged 40 to 65 years
* Absence of menstrual period for at least 2 years
* Homozygotes for the ADH1C*1 or ADH1C*2 allele of ADH1C I349V polymorphism
* Alcohol consumption ≥ 5 and ≤ 21 units/week

Exclusion Criteria:

* Smoking
* Family history of alcoholism
* History of medical or surgical events that may significantly affect the study outcome, particularly metabolic or endocrine disorders and gastrointestinal disorders
* Recent blood donation

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2006-03; Study Completion 2006-06

PRIMARY OUTCOMES:
PPAR-gamma activated gene expression

SECONDARY OUTCOMES:
Risk factors of cardiovascular disease and type 2 diabetes
Postprandial changes of HPA-axis activity

CONTACTS AND LOCATIONS:
Overall Officials: Henk FJ Hendriks, PhD., Principal Investigator — TNO

REFERENCES:
- [Derived] Joosten MM, Schrieks IC, Hendriks HF. Effect of moderate alcohol consumption on fetuin-A levels in men and women: post-hoc analyses of three open-label randomized crossover trials. Diabetol Metab Syndr. 2014 Feb 18;6(1):24. doi: 10.1186/1758-5996-6-24. PMID 24548643
- [Derived] Joosten MM, Beulens JW, Kersten S, Hendriks HF. Moderate alcohol consumption increases insulin sensitivity and ADIPOQ expression in postmenopausal women: a randomised, crossover trial. Diabetologia. 2008 Aug;51(8):1375-81. doi: 10.1007/s00125-008-1031-y. Epub 2008 May 27. PMID 18504547